CLINICAL TRIAL: NCT00570622
Title: Effect of Pioglitazone on Portal and Systemic Hemodynamics in Patients With Advanced Cirrhosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Arnulf Ferlitsch, MD, Gastroenterology and Hepatology, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIRRPIO
Record Dates: First submitted 2007-12-10; First posted 2007-12-11 (Estimated); Last update posted 2008-11-25 (Estimated); Status verified 2008-11

CONDITIONS: Cirrhosis; Ascites; Portal Hypertension
Keywords: Cirrhosis; oxidative stress; pioglitazone
MeSH Terms: conditions — Fibrosis; Ascites; Hypertension, Portal | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Patients receive 60mg of pioglitazone once a day orally for 9 days
  Interventions: Drug: Pioglitazone
- 2 (Placebo Comparator): Patients receive Placebo orally once a day for 9 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pioglitazone — Patients receive 60mg of pioglitazone once a day orally for 9 days
  Arms: 1
Drug: Placebo — Patients receive placebo once a day orally for 9 days
  Arms: 2

SUMMARY:
The purpose of this study is to investigate the response to pioglitazone on the hepatic venous pressure gradient and peripheral vascular responsiveness to vasoconstrictors in patients with advanced (Child´s Grade B or C) cirrhosis.

DETAILED DESCRIPTION:
Cirrhotic liver disease is associated with portal hypertension including elevated portal pressure as well as hyperdynamic circulation and low peripheral vascular resistance. Endothelial nitric (NO) release is impaired in liver microvasculature, upregulation of eNOS activity in the cirrhotic liver may constitute a new strategy to correct the increased hepatic vascular tone in these patients. In contrary to this impaired endothelium-dependent relaxation (endothelial dysfunction) and NO deficiency in the cirrhotic liver, systemic and splanchnic circulation of cirrhotic patients is characterized by increased vascular tone and hyporesponsiveness to vasoconstrictors. In addition to increasing insulin sensitivity, thiazolidinediones, like pioglitazone decrease oxidative stress and inflammation and improve endothelial function. In a randomized controlled, parallel group double-blind study 20 Patients with advanced (Child´s Grade B or C) liver cirrhosis will receive pioglitazone or placebo for nine days. Portal hemodynamics and forearm blood flow response will be measured at baseline and after pioglitazone/placebo to investigate the effect of pioglitazone in these group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis, grade B or C (Child-Pugh score)

Exclusion Criteria:

* History of hypersensitivity to the trial drugs and contrast agent or to drugs with a similar chemical structure
* Treatment with vasoactive or non-steroidal anti-inflammatory drugs or systemic antibiotics one week before the study
* Exclusion criteria for hepatic hemodynamic investigation
* Cardiac, renal or respiratory failure
* Previous surgical or transjugular intrahepatic portosystemic shunt
* Insulin-dependent diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-12; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
portal and systemic hemodynamic parameters | 9 days

SECONDARY OUTCOMES:
markers of oxidative stress (malondialdehyde) | 9 days

CONTACTS AND LOCATIONS:
Overall Officials: Arnulf Ferlitsch, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Internal Medicine III, Gastroenterology and Hepatology, Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Background] Ferlitsch A, Pleiner J, Mittermayer F, Schaller G, Homoncik M, Peck-Radosavljevic M, Wolzt M. Vasoconstrictor hyporeactivity can be reversed by antioxidants in patients with advanced alcoholic cirrhosis of the liver and ascites. Crit Care Med. 2005 Sep;33(9):2028-33. doi: 10.1097/01.ccm.0000178173.27923.eb. PMID 16148476